CLINICAL TRIAL: NCT06970106
Title: A Phase 1b Open-Label, Randomized, Single Dose and Repeat Dose Study to Evaluate the Single and Repeat Dose Safety and Tolerability of Intravitreally Administered PYC-001 in Participants With Confirmed OPA1 Mutation-Associated Autosomal Dominant Optic Atrophy
Brief Title: Safety of Single and Repeat Dose of PYC-001 Eye Injections in People With Autosomal Dominant Optic Atrophy
Acronym: PYC-001-CL-102
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PYC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PYC-001-CL-102
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: OPA1 Gene Mutation; Autosomal Dominant Optic Atrophy; Hereditary Optic Atrophies; Kjer Optic Atrophy
MeSH Terms: conditions — Optic Atrophy, Autosomal Dominant; Optic Atrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1: Single Dose of 60ug (Experimental): A single dose of 60ug of PYC-001 administered intravitreally
  Interventions: Drug: PYC-001
- Cohort 2: 10ug of PYC-001, 8 weeks (Experimental): 3 doses of 10ug PYC-001, administered intravitreally in 8 weeks interval
  Interventions: Drug: PYC-001
- Cohort 3: 10ug of PYC-001, 12 weeks (Experimental): 3 doses of 10ug PYC-001, administered intravitreally in 12 weeks interval
  Interventions: Drug: PYC-001
- Cohort 4: 30ug of PYC-001, 8 weeks (Experimental): 3 doses of 30ug PYC-001, administered intravitreally in 8 weeks interval
  Interventions: Drug: PYC-001
- Cohort 5: 30ug of PYC-001, 12 weeks (Experimental): 3 doses of 30ug PYC-001, administered intravitreally in 12 weeks interval
  Interventions: Drug: PYC-001
- Cohort 6: 60ug of PYC-001, 8 weeks (Experimental): Following SRC, Single dose participant can continue to receive 3 doses of 60ug PYC-001, administered intravitreally at 8 weeks interval
  Interventions: Drug: PYC-001
- Cohort 7: 60ug of PYC-001, 12 weeks (Experimental): Following SRC, Single dose participant can continue to receive 3 doses of 60ug PYC-001, administered intravitreally at 12 weeks interval
  Interventions: Drug: PYC-001

INTERVENTIONS:
Drug: PYC-001 — PYC-001 is a peptide-phosphorodiamidate morpholino oligonucleotide administered intravitreally

SUMMARY:
This study aims to gather safety data and determine the optimal dosing regimen for PYC-001 in participants with confirmed OPA1 mutation-associated ADOA. Approximately 21 participants from across UK and Australia are expected to be enrolled, depending on safety review committee (SRC) throughout the course of the study.

Participants may be assigned to any of the following:

1. A single 60ug dose of PYC-001
2. Three doses of 10ug PYC-001 at an interval of 8 weeks
3. Three doses of 10ug PYC-001 at an interval of 12 weeks
4. Three doses of 30ug PYC-001 at an interval of 8 weeks
5. Three doses of 30ug PYC-001 at an interval of 12 weeks

   Following completion of the 4 week safety review of the single 60ug of PYC-001 cohort, and if the 60 μg dose level is deemed safe by the SRC, the following cohorts will also be available:
6. Three doses of 60ug PYC-001 at an interval of 8 weeks
7. Three doses of 60ug PYC-001 at an interval of 12 weeks

DETAILED DESCRIPTION:
This is a phase 1b open-label, randomized, single and repeat dose study to evaluate the safety and tolerability of IVT administered PYC-001 in participants with confirmed OPA1 mutation-associated ADOA.

The primary objective of this study is to gather safety data and determine the optimal dosing regimen for PYC-001.

The exploratory objectives of this study include evaluating the ocular structural and functional changes following multiple doses of IVT administered PYC-001. The PK profile of PYC-001 following multiple doses will also be assessed.

In this open-label study, PYC-001 will be injected in a single eye and ocular safety will be assessed in both eyes. Approximately 21 participants are expected to enroll and complete this study; the number of enrolled participants may vary and will be driven by decisions made by the safety review committee (SRC) throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent before any study-related activity is carried out and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects;
2. Adult males and females, aged 18 years and above at screening;
3. Body mass index ≥18.0 and ≤35.0 kg/m2
4. Have a recent (within five years) genetic diagnosis of OPA1 mutation-associated (haploinsufficiency) ADOA and/or confirmed diagnosis during pre-screening or screening, as determined by the PI. In case of complex mutation profile, eligibility will be determined in consultation with the Sponsor. Rollover participants are exempt from this criterion as their genetic diagnosis was confirmed in PYC-001-101;
5. Treatment naïve participants with best-corrected visual acuity (BCVA) of between ≤20/40 (≤70 Early Treatment of Diabetic Retinopathy Study [ETDRS] letters) and ≥20/200 (≥35 ETDRS letters). If both eyes meet this eligibility criteria, the eye with better fixation as determined by the PI in consultation with the Sponsor will be selected as the study eye and the other eye will be designated as the fellow eye. In the event that both eyes are eligible and have adequate fixation to reliably perform all study assessments, the worse eye as determined by the physician will be taken as the study eye.

   PYC-001-101 participants are exempt from this criterion and will have the same study eye and fellow eye as determined in PYC-001-101;
6. Treatment Naïve participants (participants from PYC-001-101 are exempt from this criterion) with mild to moderate visual field loss and retinal nerve fiber layer (RNFL) loss in the study eye only as determined by the Spectralis Glaucoma Module Premium Edition (GMPE) RNFL & visual field structure function data (map), specifically the outer ring (T, TS, NS, N, NI and TI), defined as:

   1. Mild disease = RNFL abnormalities (outside normal range) in no more than one of six sectors;
   2. Moderate disease = RNFL abnormalities (outside normal range) in no more than three of six sectors;
   3. Severe disease = RNFL abnormalities (outside normal range) in four of six sectors;
   4. Advanced disease = RNFL abnormalities (outside normal range) in six of six sectors;
7. Medically healthy (in the opinion of the PI), as determined by pre-study medical history, and without clinically significant abnormalities including (assessments may be repeated at the discretion of the PI if an out-of-range value is determined to be erroneous):

   1. Physical examination without any clinically relevant findings;
   2. Systolic blood pressure (BP) in the range of 90 to 160 mmHg and diastolic BP in the range of 50 to 95 mmHg after five minutes in sitting or supine or semi-supine position;
   3. Heart rate (HR) in the range of 45 to 110 bpm after five minutes rest in sitting or supine or semi-supine position;
   4. Body temperature (tympanic), between 35.5°C and 37.7°C;
   5. No clinically significant findings in clinical chemistry, hematology, coagulation and urinalysis tests at screening .
8. Female participants must be of non-childbearing potential, i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least six weeks before the screening visit) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle stimulating hormone [FSH] level consistent with postmenopausal status, per local laboratory guidelines). Females receiving hormone replacement therapy (HRT) may be considered for inclusion if the need for HRT is for no other medical reason than to treat symptoms associated with menopause.

   If female participants are of childbearing potential, they must:
   1. Have a negative pregnancy test at the screening visit and on study Day -1;
   2. Agree not to attempt to become pregnant or donate ova from signing of the consent form until at least 130 days after final IVT dose administration of PYC-001;
   3. Agree to use adequate contraception (defined as use of a condom by the male partner combined with use of a highly effective method of contraception from one month prior to screening until at least 130 days after final IVT dose administration of PYC-001 , if not exclusively in a same-sex relationship or abstinent as a committed lifestyle.
9. Male participants must:

   1. Agree not to donate sperm from signing the consent form until at least 190 days after final IVT dose administration of PYC-001;
   2. If engaging in sexual intercourse with a female partner who could become pregnant, agree to use adequate contraception (defined as use of a condom combined with use of a highly effective method of contraception (defined in Appendix 13.1) from signing the consent form until at least 190 days after final IVT dose administration of PYC-001;
   3. If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, agree to use a condom from signing the consent form until at least 190 days after final IVT dose administration of PYC-001 and;
10. Willing and able to comply with all study assessments and protocol schedule/ restrictions

Exclusion Criteria:

1. Participant has a known allergy to PYC-001 or any of its excipients;
2. Demonstrated clinically significant co-morbidities, which, in the opinion of the PI, would interfere with the participant's ability to participate in the study and/or confound study outcomes;
3. Females who are breastfeeding or planning to breastfeed;
4. Based on recent (within five years of screening [for rollover PYC-001-101 participants, within five years of entry into PYC-001-101]) genetic testing, the participant has mutations in genes that cause ADOA, other than OPA1 (for example in case of dominant negative ADOA and ADOA Plus) or has other pathological variants that result in an ADOA-like optic atrophic phenotype or other pathologic genetic findings indicating presence of additional confounding ocular diseases based on comprehensive genetic screening. Eligibility will be determined by the PI in consultation with the Sponsor as needed;
5. Have received any prior cell or gene therapy for a retinal condition, excluding participation in study PYC-001-101;
6. Within three months prior to study Day -1, have undergone any vitreoretinal surgery (scleral buckle, pars plana vitrectomy, retrieval of a dropped nucleus or intraocular lens, radial optic neurotomy, sheathotomy, cyclodestructive procedures or multiple filtration surgeries [two or more]) or any other ocular surgery in the study eye.
7. Within three months prior to study Day -1, have placement of an Ozurdex® implant. This criterion does not apply for rollover participants from PYC-001-101;
8. Within three years prior to study Day -1, have placement of Retisert® of Iluvien® implants. This criterion does not apply for rollover participants from PYC-001-101;
9. Have ocular media opacity or poor pupillary dilation prohibiting quality ophthalmic evaluation or photography, as assessed by the PI in the study eye ;
10. Macular edema (intraretinal, sub-retinal or other fluid) in the study eye requiring treatment.
11. History of recurrent uveitis (idiopathic or immune-related) or active ocular inflammation;
12. Have used within 30 days of the Screening visit or is using any investigational drug (excluding PYC-001 from participation in PYC-001-101) or over-the-counter drug such as Idebenone, Vitamin B6, Vitamin B12, or a device which in the opinion of the PI or Sponsor could affect the optic nerve and/or influence functional vision or visual function during the study period. A decision will be made on a case-by-case basis by the PI in consultation with the Sponsor. Participation in observational studies is allowable based on PI discretion and consultation with the Sponsor's Medical Representative. Participation in PYC-001-101 is allowed;
13. Over-the-counter drugs like CoQ10 and other Nutraceutical usage will require a washout by five half-lives prior to baseline visit. Participants may need to stop taking the drug for the duration of the study based on Physician discretion and in consultation with the Medical Monitor;
14. Have a recent history (<6 months) of or current excessive recreational drug or alcohol use, in the opinion of the PI. Excessive alcohol use is defined as regular consumption of >10 standard drinks per week or >4 standard drinks per day, where one standard drink is defined as 10 grams of pure alcohol;
15. Positive alcohol breath test as assessed at screening, and on study Day -1 and study Day 1;
16. Positive urine drugs of abuse as assessed at screening and on study Day -1 and study Day 1;
17. Any retinal pathology other than ADOA or any other condition or prior therapy that in the opinion of the PI would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements;
18. Presence of illness or pathology that, per investigator, include symptoms and/or the associated treatments that can alter visual function. For example, cancers or pathology of the central nervous system, including multiple sclerosis;
19. Positive test for human immunodeficiency virus, hepatitis B or C virus;
20. Clinically significant findings in clinical chemistry, hematology, coagulation and urinalysis tests at screening, defined as:

    * Alanine transaminase (ALT) or aspartate aminotransferase (AST) >2 × upper limit of normal (ULN) or bilirubin >1.5 × ULN (unless patient has Gilbert's syndrome);
    * Estimated glomerular filtration rate <60 mL/min/1.73 m2; Australia, Version 3.0, 12 JUN 2025 44 Confidential
    * Hemoglobin A1c level ≥7.0%;
    * International normalized ratio ≥1.2;
    * Hemoglobin <10 g/dL, platelets <100,000/μL, and white blood cells within the normal range;
    * Clinically significant abnormalities in the urine analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
(Cohort 1) Adverse Events | 48 weeks
  To evaluate the safety and tolerability of a single dose of IVT administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA.
  * Incidence, type, severity and relationship of ocular TEAEs, and treatment-emergent SAEs in the study eye at Week 4 (±7 days), Week 8 (±7 days), Week 24 (±2 weeks), and Week 48 (±2 weeks).
  * Incidence, type, severity and relationship of ocular TEAEs, and treatment-emergent SAEs in the fellow eye at Week 4 (±7 days), Week 8 (±7 days), Week 24 (±2 weeks), and Week 48 (±2 weeks).
  * Incidence, type, severity and relationship of non-ocular TEAEs, and treatment-emergent SAEs at Week 4 (±7 days), Week 8 (±7 days), Week 24 (±2 weeks), and Week 48 (±2 weeks).
(Cohort 1) Heart Rate change from baseline at Week 8/Week 48 | 8 / 48 Weeks
  To evaluate the safety and tolerability of a single dose of IVT administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA.
(Cohort 1) Blood Pressure Change from baseline at Week 8/Week 48 | 8 Weeks/ 48 Weeks
  To evaluate the safety and tolerability of a single dose of IVT administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA
(Cohort 1) Tympanic temperature change from baseline at Week 8/Week 48 | 8 weeks / 48 weeks
  To evaluate the safety and tolerability of a single dose of IVT administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA
(Cohort 1) Respiratory rate change from baseline at Week 8 / Week 48 | 8 weeks / 48 weeks
  To evaluate the safety and tolerability of a single dose of IVT administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA
(Cohort 1) Change from baseline for clinical laboratory results - hematology to Week 8 / Week 48 | 8 Weeks / 48 Weeks
  Hematology Screening parameters: Hematocrit, Hemoglobin, Mean Corpuscular hemoglobin, mean corpuscular hemoglobin concentration, mean corpuscular volume, mean platelet volume, packed cell volume, platelet count, red blood cell count, reticulocyte count, white blood cell count with differential neutrophil count, eosinophil count, basophil count, lymphocyte count, monocyte count.
(Cohort 1) Change from baseline for clinical laboratory results - clinical chemistry to Week 8/Week 48 | 8 Weeks / 48 Weeks
  Clinical Chemistry screening parameters: Albumin, alkaline phosphatase, alanine aminotransferase, amylase, anion gap, aspartate aminotransferase, bicarbonate, calcium, ionized calcium, chloride, conjugated (direct) and unconjugated bilirubin, creatinine, eGFR, Creatinine kinase, Gamma glutamyl transferase, Globulin, Glucose, High density lipoprotein, Lactate dehydrogenase, Lipase, Low density lipoprotein, Magnesium, Phosphate, Potassium, Sodium, Total bilirubin, Total cholesterol, Total protein, Triglycerides, Urate, Urea
(Cohort 1) Change in coagulation - Clinical laboratory results from baseline to Week 8/Week 48 | 8 Weeks / 48 Weeks
  Coagulation screening parameters: Activated partial thromboplastin time, International normalized ratio/Prothrombin time, Fibrinogen
(Cohort 1) Change in urinalysis - Clinical laboratory results from baseline to Week 8/Week 48 | 8 Weeks / 48 Weeks
  Urinalysis screening parameters: Bilirubin, Blood, Glucose, Ketones, Leukocyte esterase, Nitrites, pH, Protein, Specific gravity, Urobilinogen
(Repeat Dose Cohorts) Adverse Events | 48 Weeks / 60 Weeks
  To evaluate the safety and tolerability of multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA. To determine optimal dose and dosing regimen for PYC-001.
  * Incidence, type, severity and relationship of ocular TEAEs, and treatment-emergent SAEs in the study eye over a 48-week (± 2 weeks) time period for 8-week dosing intervals Group, or a 60-week (± 2 weeks) time period for 12-week dosing intervals Group.
  * Incidence, type, severity and relationship of ocular TEAEs, and treatment-emergent SAEs in the fellow eye over a 48-week (± 2 weeks) time period for 8-week dosing intervals Group, or a 60-week (± 2 weeks) time period for 12-week dosing intervals Group.
  * Incidence, type, severity and relationship of non-ocular TEAEs, and treatment-emergent SAEs over a 48-week (± 2 weeks) time period for 8-week dosing intervals Group, or a 60-week (± 2 weeks) time period for 12-week dosing intervals group.
(Repeat Dose Cohorts) Heart Rate change from baseline at Week 48 / Week 60 | 48 Weeks / 60 Weeks
  To evaluate the safety and tolerability of multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA
  To determine optimal dose and dosing regimen for PYC-001.
  Week 48 for for 8-week dosing interval Group and Week 60 for 12-week dosing interval Group.
(Repeat Dose Cohorts) Blood Pressure Change from baseline at Week 48/ Week 60 | 48 Weeks / 60 Weeks
  To evaluate the safety and tolerability of multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA.
  To determine optimal dose and dosing regimen for PYC-001.
  Week 48 for 8-weeks dosing intervals Group Week 60 for 12-weeks dosing intervals Group
(Repeat Dose Cohorts) Tympanic Temperature Change from baseline at Week 48/ Week 60 | 48 Weeks / 60 Weeks
  To evaluate the safety and tolerability of multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA.
  To determine optimal dose and dosing regimen for PYC-001.
  Week 48 for 8-weeks dosing intervals Group Week 60 for 12-weeks dosing intervals Group
(Repeat Dose Cohorts) Respiratory Rate Change from baseline at Week 48/ Week 60 | 48 Weeks / 60 Weeks
  To evaluate the safety and tolerability of multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA.
  To determine optimal dose and dosing regimen for PYC-001.
  Week 48 for 8-weeks dosing intervals Group Week 60 for 12-weeks dosing intervals Group
(Repeat Dose Cohorts) Change in Clinical laboratory results - hematology from baseline at Week 48/ Week 60 | 48 Weeks / 60 Weeks
  Hematology Screening parameters: Hematocrit, Hemoglobin, Mean Corpuscular hemoglobin, mean corpuscular hemoglobin concentration, mean corpuscular volume, mean platelet volume, packed cell volume, platelet count, red blood cell count, reticulocyte count, white blood cell count with differential neutrophil count, eosinophil count, basophil count, lymphocyte count, monocyte count.
  To determine optimal dose and dosing regimen for PYC-001.
  Week 48 for 8-weeks dosing intervals Group Week 60 for 12-weeks dosing intervals Group
(Repeat Dose Cohorts) Change in Clinical laboratory results - clinical chemistry from baseline at Week 48/ Week 60 | 48 Weeks / 60 Weeks
  To evaluate the safety and tolerability of multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA.
  To determine optimal dose and dosing regimen for PYC-001.
  Week 48 for 8-weeks dosing intervals Group Week 60 for 12-weeks dosing intervals Group
(Repeat Dose Cohorts) Change in Clinical laboratory results - coagulation from baseline at Week 48/ Week 60 | 48 Weeks / 60 Weeks
  To evaluate the safety and tolerability of multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA.
  To determine optimal dose and dosing regimen for PYC-001.
  Week 48 for 8-weeks dosing intervals Group Week 60 for 12-weeks dosing intervals Group
(Repeat Dose Cohorts) Change in Clinical laboratory results - urinalysis from baseline at Week 48/ Week 60 | 48 Weeks / 60 Weeks
  To evaluate the safety and tolerability of multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated with ADOA.
  To determine optimal dose and dosing regimen for PYC-001.
  Week 48 for 8-weeks dosing intervals Group Week 60 for 12-weeks dosing intervals Group

SECONDARY OUTCOMES:
(Cohort 1) Change from Baseline for Best-corrected visual acuity letter score using Early Treatment of Diabetic Retinopathy Study | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Low contrast visual acuity | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for High contrast visual acuity | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Visual field sensitivity by photopic static perimetry | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Posterior eye health by fundus examination, using ultrawide fundoscopy | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Color vision by Hardy Rand Rittler test | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Contrast sensitivity by Pelli Robson chart | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Multifocal visual evoked potential OR Full field electroretinogram | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Retinal nerve fiber layer (RNFL) by spectral domain optical coherence tomography | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA.
  The unit for RNFL thickness is typically measured in microns or millimeters.
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Mitochondrial function test by flavoprotein fluorescence analyzer (Ocumet Beacon) | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Repeat Dose Cohort) Change from Baseline for Best-corrected visual acuity letter score using Early Treatment of Diabetic Retinopathy Study | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Low contrast visual acuity | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for High contrast visual acuity | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Visual field sensitivity by photopic static perimetry | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Posterior eye health by fundus examination, using ultrawide fundoscopy | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Color vision by Hardy Rand Rittler test | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Contrast sensitivity by Pelli Robson chart | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Multifocal visual evoked potential OR Full field electroretinogram | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Retinal nerve fiber layer (RNFL), by spectral domain optical coherence tomography | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  The unit for RNFL is usually in micrometers and sometimes in millimeters.
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Mitochondrial function test by flavoprotein fluorescence analyzer (Ocumet Beacon) | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Visual field using OLLEYES mobile device | 48 weeks / 60 Weeks
  Visual field can be measured using degrees.
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Plasma concentrations of PYC-001 following multiple dose intravitreally administered PYC-001 | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Cohort 1) Change from Baseline for Ganglion Cell Layer (GCL) thickness determined by spectral domain optical coherence tomography | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  The unit for Ganglion Cell Layer thickness is usually in micrometers.
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Cohort 1) Change from Baseline for Bruch's membrane opening (BMO) disc size as determined by spectral domain optical coherence tomography | 48 weeks
  To evaluate ocular structural and functional changes with single doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 4, Week 8, Week 12, Week 24, and Week 48
(Repeat Dose Cohort) Change from Baseline for Ganglion Cell Layer (GCL) thickness determined by Spectral domain optical coherence tomography | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  The unit for GCL thickness is usually in micrometers.
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for Bruch's membrane opening (BMO) disc size, as determined by spectral domain optical coherence tomography | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for visual acuity using OLLEYES mobile device | 48 weeks / 60 Weeks
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for contrast sensitivity using OLLEYES mobile device | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group
(Repeat Dose Cohort) Change from Baseline for color vision using OLLEYES mobile device | 48 weeks / 60 Weeks
  To evaluate ocular structural and functional changes with multiple doses of intravitreally administered PYC-001 in participants with confirmed OPA1 mutation associated ADOA
  Change from baseline at Week 48 for 8-weeks dosing interval Group and Week 60 for 12-weeks dosing interval Group

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Save Sight Institute - Sydney Eye Hospital, Sydney, New South Wales
  - Cerulea Clinical Trials, East Melbourne
- Retina Specialists, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No